CLINICAL TRIAL: NCT04926727
Title: Prevalence And Burden Of Nausea And Vomiting In Pregnant Women. An Italian Survey (PURITY)
Brief Title: Prevalence And Burden Of Nausea And Vomiting In Pregnant Women
Acronym: PURITY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Italfarmaco (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: OPITA/0120/SU
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Nausea Gravidarum; Vomiting of Pregnancy
Keywords: Nausea of Pregnancy; Vomiting of Pregnancy; Survey; Italy; Nuperal®
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: 600 Pregnant women between the 18th and 22nd week.
  * 200 from Northern Italy;
  * 200 from Central Italy;
  * 200 from Southern Italy and the Islands.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Observational study

SUMMARY:
On February 25th, 2019, ITALFARMACO launched Nuperal® in Italy, an association of doxylamine succinate and pyridoxine hydrochloride authorized by AIFA for the symptomatic treatment of nausea and vomiting in pregnancy (NVP). This drug is also recommended as first choice drug therapy by the American College of Obstetricians and Gynecologists (ACOG) Guidelines and is supported by extensive international literature.

Numerous epidemiological researches conducted in the US and Norway have highlighted the extent of vomiting and pregnant nausea. Unfortunately to date, there are no information on the prevalence of this phenomenon in Italy, on its impact on women's lives and on the interaction between woman and gynecologists.

The research hypothesis of the present survey is that, using a representative sample of pregnant women in Italy, it will be possible to identify the prevalence and weight of nausea and vomiting symptoms during pregnancy in this country. The study is an open, non-comparative, multicenter survey and the aim is to evaluate the prevalence and weight that the symptoms of nausea and vomiting have in pregnant women in Italy.

The study population will include 600 women found during weeks 18-22 of pregnancy who will arrive at the three sites or will contact the Investigators after the Ethics Committee (EC) approval.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian women in physiological pregnancy and between the 18th and 22nd week (time of morphological ultrasound).
* Women able to communicate adequately with the interviewer and understand the questionnaires.
* Women able to understand and who can provide valid informed consent to the Survey.

Exclusion Criteria:

* Twin pregnancy.
* Medically assisted procreation (MAP)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Caucasian women in physiological pregnancy between the 18th and 22nd week (time of morphological ultrasound).
Study Population: Pregnant women between the 18th and 22nd week. Inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
NVP prevalence. | 18 to 22 weeks
  Nausea, vomiting pregnancy prevalence
Percentage of cases based on PUQE | 18 to 22 weeks
  Percentage of mild, medium and severe cases based on PUQE.
NVP related questions | 18 to 22 weeks
  Percentage of answer allocation to Nausea Vomiting Pregnancy related questions
Mean and SD of onset for each symptom and its duration | 18 to 22 weeks
  Mean and Standard Deviation of onset for each symptom and its duration
Correlations between demographic data and the presence of symptoms | 18 to 22 weeks
  Correlations between demographic data (age, first pregnancy status, multiparity, geographical origin, type of work and educational qualification) and the presence of symptoms and their severity.
Correlation with the use of both therapies | 18 to 22 weeks
  Correlation of the use of non-pharmacological, pharmacological or both therapies with the severity of the symptoms during pregnancy and with the possible outcomes.
Correlation between severity of symptoms and consequences on women's personal life. | 18 to 22 weeks
  Correlation between severity of symptoms and consequences on women's personal life (family, work, etc.).
Number of cases with hospitalization | 18 to 22 weeks
  Number of cases with hospitalization in relation to total and severity of symptoms (PUQE).
Correlation between symptoms in pregnancy and outcomes based on data from the post pregnancy questionnaire | 18 to 22 weeks
  Correlation between symptoms in pregnancy (and relative severity) and outcomes based on data from the post pregnancy questionnaire (weight of new-born, gestational age at birth and any complications).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Policlinico di Napoli - Università di Napoli "Federico II", Napoli, Corso Umberto I 40
  - P.O. SS.ma Annunziata di Chieti della ASL di Chieti, Chieti, Via Dei Vestini
  - Ospedale dei Bambini "Vittore Buzzi", Milan, Via Lodovico Castelvetro, 32

IPD SHARING:
Plan to Share IPD: Undecided